CLINICAL TRIAL: NCT00243243
Title: Effect of Recombinant Coagulation Factor VIIa on Peri-operative Blood Loss in Patients Undergoing Major Burn Excision and Grafting
Brief Title: Effect of rFVIIa on Peri-operative Blood Loss in Patients Undergoing Major Burn
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-05-027
Record Dates: First submitted 2005-10-19; First posted 2005-10-21 (Estimated); Results first posted 2013-03-06 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Burns
Keywords: Burns
MeSH Terms: conditions — Burns | interventions — recombinant FVIIa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rFVIIa (Experimental): intravenous administration of rFVIIa (Novoseven; 90 micrograms/kg, IV push, given at start of first surgical incision and again at 1 hr after start of surgery)
  Interventions: Drug: Recombinant Factor VIIa
- Control (Placebo Comparator): intravenous administration of placebo (sterile water, IV push, given at first surgical incision and again at 1 hr after start of surgery)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Recombinant Factor VIIa — intravenous infusion of Factor VIIa
  Arms: rFVIIa
Drug: Placebo — intravenous infusion of placebo (sterile water)
  Arms: Control

SUMMARY:
The purpose of the study is to see if a medication (Recombinant Coagulation Factor VIIa or NovoSeven), normally used to stop bleeding in persons with a bleeding disorder, will lower the amount of blood lost during burn surgery.

DETAILED DESCRIPTION:
To identify the clinical use for Factor VIIa in the operating room to reduce blood loss and blood transfusion , determine the Recombinant Factor VIIa (rFVIIa) pharmacokinetics in burned patients, determine if fFVIIa should be used to reduce peri-operative blood loss in patients undergoing excision greater than or equal to 20 percent of the total body surface area, determine the efficacy of the drug in burned patients undergoing excision of burn wounds.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Burn wounds
* 18-65 years of age
* Scheduled excision of burn wound of at least 20 percent TBSA

Exclusion Criteria:

* Age greater than 65 years
* History of blood coagulation disorders
* Taking anti-coagulation medication
* Contraindication for heparin therapy
* Pregnant or nursing females
* Unstable angina
* MI within the last 6 months
* Recent of diagnosis of DVT, stroke within the last 6 months
* Renal failure requiring dialysis or creatinine clearance less than 25 ml/min
* Religious prohibition to blood transfusion
* Have received rFVIIa during current hospitalization
* Previous enrollment in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-01; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myung S Park, MD, Principal Investigator — United States Army Institute of Surgical Research
Locations (1):
- United States Army Institute of Surgical Research, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deveras RA, Kessler CM. Reversal of warfarin-induced excessive anticoagulation with recombinant human factor VIIa concentrate. Ann Intern Med. 2002 Dec 3;137(11):884-8. doi: 10.7326/0003-4819-137-11-200212030-00009. PMID 12458988

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with greater than 20% TBSA burn scheduled for excision and grafting will be randomized in the operating room.
Pre-assignment Details: If the excision and grafting was not the first for the patient.
Groups:
- Experimental: Recombinant Factor VIIa : intravenous infusion of Factor VIIa
- Control- Placebo: Intravenous infusion of a placebo
Period: Overall Study
Arm/Group | Experimental | Control- Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (8.33) | 28.8 (10.24) | 29.1 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Blood Components Transfused During and up to 24 Hours Post Operatively
Time Frame: 24 hours
Measure: Number; unit: units of blood components
Arm/Group | Experimental | Control- Placebo
Number analyzed (Participants) | 10 | 10
units of blood components
  Units of PRBC | 68.9 | 87.2
  Units of cryoprecipitate | 0 | 4.1
  Units of platelets | 1.02 | 6.45
  Units of fresh frozen plasma | 13.02 | 33.44

ADVERSE EVENTS:
Arm/Group | Experimental | Control
Serious Adverse Events (participants affected / at risk) | 7/10 | 5/10
Other Adverse Events (participants affected / at risk) | 7/10 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=10) | Control (N=10)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Sepsis (Immune system disorders) | 2 (2) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 3 (3)
Muscle Necrosis (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1)
Bacteremia (Immune system disorders) | 1 (3) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
MI (Cardiac disorders) | 1 (1) | 1 (1)
Vascular Disorders (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=10) | Control (N=10)
Infection (Immune system disorders) | 7 (17) | 5 (9)
Rule Out Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Decreased Oxygen Saturation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Renal Insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotension (Blood and lymphatic system disorders) | 2 (2) | 2 (3)
Liver Injury (Hepatobiliary disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper Extremity Edema (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes